CLINICAL TRIAL: NCT03972280
Title: A Multicenter, Open-label, 2-regimen, Repeat-dose Study to Assess the Safety and Pharmacokinetics of Intravenous CSL324 in Subjects With Hidradenitis Suppurativa and Palmoplantar Pustulosis
Brief Title: Safety and Pharmacokinetics of Repeat Doses of CSL324 in Subjects With Hidradenitis Suppurativa and Palmoplantar Pustulosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSL324_1002; 2018-002871-17 (EudraCT Number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Hidradenitis Suppurativa; Palmoplantar Pustulosis
MeSH Terms: conditions — Hidradenitis Suppurativa; Psoriasis | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (HS) (Experimental): Dose 1 of recombinant anti-G-CSF receptor monoclonal antibody administered intravenously to subjects with HS
  Interventions: Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody
- Dose Level 1 (PPP) (Experimental): Dose 1 of recombinant anti-G-CSF receptor monoclonal antibody administered intravenously to subjects with PPP
  Interventions: Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody
- Dose Level 1 (Total) (Experimental): Dose 1 of recombinant anti-G-CSF receptor monoclonal antibody administered intravenously to subjects with HS or PPP
  Interventions: Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody
- Dose Level 2 (HS) (Experimental): Dose 2 of recombinant anti-G-CSF receptor monoclonal antibody administered intravenously to subjects with HS
  Interventions: Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody
- Dose Level 2 (PPP) (Experimental): Dose 2 of recombinant anti-G-CSF receptor monoclonal antibody administered intravenously to subjects with PPP
  Interventions: Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody
- Dose Level 2 (Total) (Experimental): Dose 2 of recombinant anti-G-CSF receptor monoclonal antibody administered intravenously to subjects with HS or PPP
  Interventions: Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody

INTERVENTIONS:
Biological: Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody — Recombinant anti-G-CSF receptor monoclonal antibody is a preservative-free, sterile liquid formulation that is suitable for intravenous infusion
  Other Names: CSL324

SUMMARY:
Study CSL324_1002 will investigate the safety and pharmacokinetics of repeat doses of CSL324 in subjects with hidradenitis suppurativa and palmoplantar pustulosis. CSL324 is a novel, recombinant therapy that may treat diseases caused by increased numbers of neutrophils at sites of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 75 years of age, inclusive
* Confirmed clinical diagnosis of moderate to severe HS as per International Hidradenitis Suppurativa Severity Score System (IHS4) guidelines (ie, IHS4 ≥ 4)
* PPP differentiated from other forms of pustulosis
* Psoriasis with a Palmoplantar Pustulosis Psoriasis Area and Severity Index (ppPASI) score of ≥ 12.
* Subjects with HS only: inadequate response to at least a 3-month (90 days) trial of oral antibiotics for treatment of HS
* Subjects with PPP only: confirmed clinical diagnosis of PPP at least 6 months before Screening and inadequate response to topical therapy, phototherapy, and / or previous systemic therapy for the treatment of PPP

Exclusion Criteria:

* Treatment with any medications and therapies not permitted during the study.
* History of myeloproliferative disease.
* Malignancy within 5 years at Screening with the exception of nonmelanoma skin cancer, carcinoma in situ, or prostate cancer not requiring treatment.
* Current, or a recent clinically significant history of, uncontrolled renal, hepatic(including currently active hepatitis B virus and / or hepatitis C virus), hematologic, endocrine, pulmonary, psychiatric, or cardiac disease, assessed as potentially having an effect on study outcomes as determined by the Investigator and / or Sponsor.
* Congenital or acquired immunosuppressive condition(s), including human immunodeficiency virus infection.
* Clinical signs of active infection and / or fever > 38°C during the 7 days before Day 1.
* Clinically significant abnormalities on physical examination, ECG, or laboratory assessments, or neutropenia (defined as absolute neutrophil count < 2.0 × 109/L) at Screening.
* Subjects with PPP only: concurrent psoriasis vulgaris (not including scaly scalp and / or ears).
* Subjects with HS only: > 20 draining fistulas."

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 24 weeks
TEAEs by severity | Up to 24 weeks
TEAEs by casuality | Up to 24 weeks
Incidence of adverse events of special interest (AESIs): Grade 3 and 4 neutropenia | Up to 24 weeks
AESIs: Grade 3 and 4 neutropenia by causality | Up to 24 weeks
Incidence of AESIs: Grade 3 and 4 infection | Up to 24 weeks
AESIs: Grade 3 and 4 infection by causality | Up to 24 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of CSL324 in serum for the first dose administered | Up to 22 days after dose
Time to maximum concentration (Tmax) of CSL324 in serum for the first dose administered | Up to 22 days after dose
Area under the concentration-time curve during a dosing interval (AUCtau) of CSL324 in serum for the first dose administered | Up to 22 days after dose
Cmax of CSL324 in serum for the last dose administered | Up to 22 days after dose
Tmax of CSL324 in serum for the last dose administered | Up to 84 days after dose
AUCtau of CSL324 in serum for the last dose administered | Up to 22 days after dose
Half life (t½) of CSL324 in serum for the last dose administered | Up to 84 days after dose
Total systemic clearance (CLtot) after intravenous dosing of CSL324 in serum for the last dose administered | Up to 22 days after dose
Volume of distribution after intravenous dosing during the terminal elimination phase ( Vz) of CSL324 in serum for the last dose administered | Up to 22 days after dose
Ctrough of CSL324 for each dose of CSL324 administered | Up to 22 days after each dose
Accumulation ratio for AUCtau (ratio between AUCtau of the last dose and of the first dose) and accumulation ratio for Cmax (ratio between Cmax of the last dose and of the first dose) | Up to 22 days after each dose
Presence of anti-CSL324 antibodies in serum | Up to 168 days

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (4):
  - Holdsworth House Medical Practice, Darlinghurst
  - Fremantle Dermatology, Fremantle
  - The Royal Melbourne Hospital, Parkville
  - Westmead Hospital, Westmead
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Hellerup
  - Zealand University Hospital, Roskilde
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - St. Josef Hospital, Bochum
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Carl Gustav Carus, Dresden

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.